CLINICAL TRIAL: NCT03893201
Title: Multi-Centre Registry to Investigate the Efficacy and Safety of Venaseal Endovenous Ablation for Varicose Veins in Singapore
Brief Title: A Singapore Venaseal Real World Post-Market Evaluation Study
Acronym: ASVS
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/2087
Record Dates: First submitted 2019-03-04; First posted 2019-03-28 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Varicose Veins; Venous Reflux; Chronic Venous Insufficiency
Keywords: Endovenous Ablation
MeSH Terms: conditions — Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venaseal: Patients that have undergone venaseal
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires to assess quality of life

SUMMARY:
The study aims to assess the efficacy of VenaSeal™ Closure System (VCS) for the treatment of lower extremity superficial truncal veins in a real-world clinical setting, in a multi-racial Asian population in Singapore.

DETAILED DESCRIPTION:
The purpose of the ASVS study is to investigate the performance of cyanoacrylate glue closure (CAC) in a real-world post market evaluation setting in which multiple incompetent superficial saphenous truncal veins - namely (great saphenous vein (GSV), short saphenous vein (SSV), anterior accessory saphenous vein (AASV) - will be treated at the same setting, and compression stockings will not be used postoperatively. Unlike previous studies, the inclusion criteria for this study will be liberalized, and veins up to 12mm in diameter will be treated. As such, ASVS will be the first published prospective trial conducted in Asia on a predominantly Asian cohort of patients to report on the performance of CAC for incompetent GSV and non-GSV trunks. This study specifically focuses on the initial technical outcomes, safety, anatomical occlusion and patient experience with CAC applied with broader inclusion of patients than previous trials.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years old and able to understand the requirements of the study and to provide informed consent
* C2 - C5 symptomatic veins / Chronic Venous Insufficiency
* Symptomatic primary GSV, SSV or AASV incompetence, with reflux > 0.5 seconds on colour Duplex, including one or more of the following symptoms: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling
* Patients who had GSV, SSV or AASV diameters of 3mm to 12mm in the standing position

Exclusion Criteria:

* Current DVT or history of DVT
* Recurrent varicose veins
* Pregnant patients
* Arterial Disease (ABPI<0.8)
* Sepsis
* Patients who are unwilling to participate
* Inability or unwillingness to complete questionnaires
* Adverse reaction to sclerosant or cyanoacrylate
* GSV, SSV or AASV severely tortuous
* Life expectancy < 1 year
* Active treatment for malignancy other than non-melanoma skin cancer
* Current, regular use of systemic anticoagulation (e.g. warfarin, heparin)
* Daily use of narcotic analgesia or NSAIDS to control pain associated with venous disease

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will be undergoing Venaseal™ as treatment for their varicose veins / chronic venous insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Technical Success at time of procedure | Immediately post-op
  Occlusion of treated vein post-procedure
Change in anatomy of treated vessel | 2 weeks, 3 months, 6 months and 12 months post-procedure
  Anatomical Success as measured at each timepoint using ultrasound to ensure no re-opening of treated vessel

SECONDARY OUTCOMES:
Quality of Life Score using the EQ-5D questionnaire | Baseline, 2 weeks, 3 months, 6 months and 12 months post-operation
  EQ5D is used to assess quality of life based on Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime.
Quality of Life Score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | Baseline, 2 weeks, 3 months, 6 months and 12 months post-operation
  CIVIQ is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging for 0 to 100 - the higher the value, the poorer the quality of life.
Quality of Life score using the Aberdeen Varicose Vein Questionnaire (AVVQ) | Baseline, 2 weeks, 3 months, 6 months and 12 months post-operation
  To measure health status of varicose veins patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life
Clinical Change usin Venous Clinical Severity Score (VCSS) | Baseline, 2 weeks, 3 months, 6 months and 12 months post-operation
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (mild), 2 (moderate), 3 (severe).
Pain Score | First 10 days post-operation
  Using a numerical rating scale, which ranges from 0 (no pain) to 10 (severe pain)
Time taken to return to work and normal activities | 10 days post-op
Occlusion rates | 2 weeks, 3 months, 6 months and 12 months post-operation
  Duplex ultrasound performed at specific timepoints to ensure that treated vein is occluded
Patient satisfaction with treatment | 2 weeks, 3 months, 6 months and 12 months post-procedure
  A short survey to assess patient satisfaction and if there are any observed improvement in terms of appearance and symptoms post-procedure.
Cost Effectiveness of the intervention | 12 months post-procedure
  To evaluate the cost involved with procedure performed

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nesbitt C, Bedenis R, Bhattacharya V, Stansby G. Endovenous ablation (radiofrequency and laser) and foam sclerotherapy versus open surgery for great saphenous vein varices. Cochrane Database Syst Rev. 2014 Jul 30;(7):CD005624. doi: 10.1002/14651858.CD005624.pub3. PMID 25075589
- [Background] Siribumrungwong B, Noorit P, Wilasrusmee C, Attia J, Thakkinstian A. A systematic review and meta-analysis of randomised controlled trials comparing endovenous ablation and surgical intervention in patients with varicose vein. Eur J Vasc Endovasc Surg. 2012 Aug;44(2):214-23. doi: 10.1016/j.ejvs.2012.05.017. Epub 2012 Jun 15. PMID 22705163
- [Background] Darwood RJ, Theivacumar N, Dellagrammaticas D, Mavor AI, Gough MJ. Randomized clinical trial comparing endovenous laser ablation with surgery for the treatment of primary great saphenous varicose veins. Br J Surg. 2008 Mar;95(3):294-301. doi: 10.1002/bjs.6101. PMID 18278775
- [Background] Rasmussen LH, Lawaetz M, Bjoern L, Vennits B, Blemings A, Eklof B. Randomized clinical trial comparing endovenous laser ablation, radiofrequency ablation, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1079-87. doi: 10.1002/bjs.7555. PMID 21725957
- [Background] Marsden G, Perry M, Kelley K, Davies AH; Guideline Development Group. Diagnosis and management of varicose veins in the legs: summary of NICE guidance. BMJ. 2013 Jul 24;347:f4279. doi: 10.1136/bmj.f4279. No abstract available. PMID 23884969
- [Background] Shepherd AC, Gohel MS, Brown LC, Metcalfe MJ, Hamish M, Davies AH. Randomized clinical trial of VNUS ClosureFAST radiofrequency ablation versus laser for varicose veins. Br J Surg. 2010 Jun;97(6):810-8. doi: 10.1002/bjs.7091. PMID 20473992
- [Background] Rabe E, Otto J, Schliephake D, Pannier F. Efficacy and safety of great saphenous vein sclerotherapy using standardised polidocanol foam (ESAF): a randomised controlled multicentre clinical trial. Eur J Vasc Endovasc Surg. 2008 Feb;35(2):238-45. doi: 10.1016/j.ejvs.2007.09.006. Epub 2007 Nov 7. PMID 17988905
- [Background] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Background] Tang TY, Kam JW, Gaunt ME. ClariVein(R) - Early results from a large single-centre series of mechanochemical endovenous ablation for varicose veins. Phlebology. 2017 Feb;32(1):6-12. doi: 10.1177/0268355516630154. Epub 2016 Jul 9. PMID 26908638
- [Background] Vanlangenhove P, De Keukeleire K, Everaert K, Van Maele G, Defreyne L. Efficacy and safety of two different n-butyl-2-cyanoacrylates for the embolization of varicoceles: a prospective, randomized, blinded study. Cardiovasc Intervent Radiol. 2012 Jun;35(3):598-606. doi: 10.1007/s00270-011-0188-9. Epub 2011 Jun 3. PMID 21638147
- [Background] Brothers MF, Kaufmann JC, Fox AJ, Deveikis JP. n-Butyl 2-cyanoacrylate--substitute for IBCA in interventional neuroradiology: histopathologic and polymerization time studies. AJNR Am J Neuroradiol. 1989 Jul-Aug;10(4):777-86. PMID 2505505
- [Derived] Tang TY, Yap CJQ, Chan SL, Soon SXY, Khoo VBX, Choke E, Chong TT. 3-year clinical outcomes of A Singapore VenaSeal real world post-market evaluation Study (ASVS) for varicose vein ablation. CVIR Endovasc. 2024 Apr 27;7(1):41. doi: 10.1186/s42155-024-00452-8. PMID 38676860
- [Derived] Tang TY, Yap CJQ, Chan SL, Soon SXY, Yap HY, Lee SQW, Choke ETC, Chong TT. Early results of an Asian prospective multicenter VenaSeal real-world postmarket evaluation to investigate the efficacy and safety of cyanoacrylate endovenous ablation for varicose veins. J Vasc Surg Venous Lymphat Disord. 2021 Mar;9(2):335-345.e2. doi: 10.1016/j.jvsv.2020.03.020. Epub 2020 May 7. PMID 32387378